CLINICAL TRIAL: NCT02103881
Title: A Double Blinded Randomized Trial of Ketamine Versus Haloperidol for Severe Prehospital Agitation
Brief Title: Ketamine Versus Haloperidol for Severe Agitation Outside the Hospital
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSR #13-3682
Record Dates: First submitted 2014-02-20; First posted 2014-04-04 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Agitation
Keywords: Agitation; Ketamine; Haloperidol; Emergency Medical Services; Feeling of restlessness; Increased motor activity
MeSH Terms: conditions — Psychomotor Agitation | interventions — Ketamine; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Ketamine (Experimental): Patients enrolled in this arm will be given 500 mg of intramuscular ketamine for their severe agitation they experience in the prehospital environment.
  Interventions: Drug: Ketamine
- Haloperidol (Experimental): Patients enrolled in this arm will be given 10 mg of intramuscular haloperidol for their severe agitation they experience in the prehospital environment.
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Drug: Ketamine — 500 mg of intramuscular ketamine for severe pre-hospital agitation
  Other Names: Ketalar
  Arms: Ketamine
Drug: Haloperidol — Haloperidol 10 mg intramuscular for severe prehospital agitation.
  Other Names: Haldol
  Arms: Haloperidol

SUMMARY:
This research study is being done to find out if one of two drugs, ketamine or haloperidol, is better for treating agitation. Agitation is a state of extreme emotional disturbance where patients can become physically aggressive or violent, endangering themselves and those who are caring for them. Often chemical substances or severe mental illness is involved in this level of agitation. Specifically, the investigators are interested in studying agitation that is treated in the prehospital setting by paramedics. This study's hypothesis is that ketamine is superior to haloperidol for treatment of agitation in the prehospital environment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of severe agitation in the prehospital environment

Exclusion Criteria:

* Prisoners
* Persons known to be younger than 18 years old
* Persons suspected to be younger than 18 years old
* Obviously gravid women
* Persons with profound agitation
* Persons who are unable to be transported to the treating facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Time from injection of drug to adequate sedation, defined as a score of 0 or less on the AMSS. | 2 hours
  The Altered Mental Status Scale (AMSS) is an integral ordinal scale evaluating both agitation and sedation with scores from -4 to +4. It was developed at our institution and has been internally and externally validated. This scale is a modified version of the Behavioral Activity Rating Scale with additional data points from the Observer's Assessment of Alertness Scale. Effectiveness of sedation will be defined as an AMS score less than or equal to 0.
  AMSS will be determined by the treating paramedic, who will undergo training as a research associate prior to commencement of the study. Participants will be followed for the duration of agitation, an expected average of 2 hours.

SECONDARY OUTCOMES:
Number of participants intubated. | 2 hours
  Participants will be followed for the duration of agitation, an expected average of 2 hours. Enrolling paramedics or research associates in the Emergency Department will record if the patient is intubated.
venous pH | at one minutes and ten minutes post sedation
  Venous blood will be drawn at one and ten minutes post sedation and assessed using point-of-care testing for pH. Enrolling paramedics or research associates in the Emergency Department will record the data.
serum potassium | at one minute and ten minutes post sedation
  Venous blood will be drawn at one and ten minutes post sedation and assessed using point-of-care testing for potassium concentration. Enrolling paramedics or research associates in the Emergency Department will record the data.
Total time the participant is a patient in the Emergency Department. | 2 hours
  Participants will be followed for the duration of agitation, an expected average of 2 hours. Enrolling paramedics or research associates in the Emergency Department will record both the time the patient arrives in the Emergency Department, and when they leave the Emergency Department.
Number of patients admitted versus number of patients discharged. | 2 hours
  Participants will be followed for the duration of agitation, an expected average of 2 hours. Enrolling paramedics or research associates in the Emergency Department will record if the patient is admitted or discharged.
venous lactate | at one minute and ten minutes post sedation
  Venous blood will be drawn at one and ten minutes post sedation and assessed using point-of-care testing for lactate concentration. Enrolling paramedics or research associates in the Emergency Department will record the data.
Number of patients experiencing laryngospasm. | 2 hours
  Participants will be followed for the duration of agitation, an expected average of 2 hours. Enrolling paramedics or research associates in the Emergency Department will record if laryngospasm occurs.
Number of patients experiencing dystonia. | 2 hours
  Participants will be followed for the duration of agitation, an expected average of 2 hours.Enrolling paramedics or research associates in the Emergency Department will record if dystonia occurs.